CLINICAL TRIAL: NCT05687604
Title: Scalable TELeheaLth Cancer CARe: The STELLAR Program to Treat Cancer Risk Behaviors
Acronym: STELLAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Brian Hitsman, Associate Professor of Preventive Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P50CA271353 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2023-01-18 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Smoking Cessation; Physical Inactivity
MeSH Terms: conditions — Obesity; Smoking Cessation; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial with 2 parallel intervention arms. One arm will be the active treatment group, and the other an enhanced usual-care control group. Assessors will be blinded to study condition, and intervention will be behavioral.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACILITATED Program (Active Comparator): STELLAR arm participants will receive goals related to their physical activity, smoking, and/or obesity, and will be asked to meet those goals weekly/daily. Participants will also be asked to record their weight, activity, and/or cigarette smoking daily, and will complete 12 telehealth sessions with study staff across the 9 months of the study. Will have physical measures taken or extracted from the medical record at baseline, 3 months, 6 months, and 9 months.
  Interventions: Behavioral: multiple behavior change therapy
- SELF GUIDED Program (No Intervention): Patients in the EUC group will receive informational packets about their risk behaviors - obesity, physical inactivity, and/or smoking. Will have physical measures taken or extracted from the medical record at baseline, 3 months, 6 months, and 9 months

INTERVENTIONS:
Behavioral: multiple behavior change therapy — goals related to their physical activity, smoking, and/or obesity, and will be asked to meet those goals weekly/daily. Participants will also be asked to record their weight, activity, and/or cigarette smoking daily, and will complete 16 telehealth sessions with study staff across the 12 months of the study. Will have physical measures taken or extracted from the medical record at baseline, 3 months, 6 months, and 12 months.
  Arms: FACILITATED Program

SUMMARY:
The goal of this clinical trial is to improve cancer patient's health, survival, and quality of life by dispelling risk behaviors for Northwestern Memorial Health Care (NMHC) patients who are cancer survivors.

The main question[s] STELLAR aims to answer are:

* How best to combine three behavior interventions (physical activity promotion, smoking cessation, obesity treatment) into one treatment.
* Evaluate the reach of the program. We will look at the number, proportion, and representativeness of participants in terms of disease characteristics, socioeconomic status, telehealth readiness, and race/ethnicity.
* Evaluate the effects of the STELLAR program relative to enhanced usual care (information provision) on cancer risk behaviors, patient care access, care quality, and communication.

Participants will be provided goals related to their physical activity, smoking, and/or weight loss and asked to track their health behaviors via an app, excel file, or on paper. At baseline, 3 months, 6 months and 9 months into the study, participants will provide survey responses and physical measurements like height and weight. Additionally, those in the Facilitated group will complete 12 telehealth sessions with study staff to discuss progress towards their study goals.

Researchers will compare the Facilitated group to the Self Guided group to see if the Facilitated intervention group is able to reach more participants that enhances care only.

DETAILED DESCRIPTION:
The goal of this clinical trial is to decrease adverse outcomes and improve cancer patient's health, survival, and quality of life by dispelling risk behaviors for Northwestern Memorial Health Care (NMHC) patients.

The main question[s] STELLAR aims to answer are:

* How best to combine three existing effective cancer risk behavior interventions (physical activity promotion, smoking cessation, obesity treatment) into one treatment program within the existing NMHC environment.
* Evaluate the reach of the FACILITATED program. We will look at the number, proportion, and representativeness of individuals who are willing to participate in terms of disease characteristics, socioeconomic status, telehealth readiness, and race/ethnicity.
* Evaluate the effects of the FACILITATED program relative to enhanced usual care (information provision) on cancer risk behaviors, patient care access, care quality, healthcare utilization, patient-provider communication, cost and health outcomes (symptoms and quality of life).

Participants will be recruited through several channels (MyNM, direct outreach from research staff, EDW). Interested patients will then be randomly assigned to the STELLAR program arm, or Enhanced Usual Care. Participants in the STELLAR program will be enrolled for a year into the program. Participants will be provided goals related to their physical activity, smoking, and/or weight loss and asked to track their health behaviors via an app, excel file, or on paper. At baseline, 3 months, 6 months and 9 months into the study, participants will provide survey responses and physical measurements like height and weight. Additionally, those in the FACILITATED group will complete 12 telehealth sessions with study staff to discuss progress towards their study goals.

Researchers will compare the FACILITATED intervention group to the SELF GUIDED group to see if the FACILITATED intervention group is able to reach more participants that Self Guided only.

ELIGIBILITY:
Inclusion Criteria:

* Northwestern Medicine patient
* Over 18 years old
* Meet at least 1 of the following 3 criteria:
* Engage in <150 min/week of physical activity
* BMI of ≥25
* Report that they currently smoke or smoked within the last year
* Diagnosed with any cancer (except non-melanoma skin)
* Ability to attend telehealth visits either via landline, cell phone, smartphone, tablet, laptop, or desktop computer
* 3 months post curative intent treatment if BMI of ≥25 or engage in <150 min/week of physical activity
* Post curative intent treatment if they currently smoke or smoked within the last year

Exclusion Criteria:

* Currently in another dietary, weight loss, smoking cessation (including cessation pharmacotherapy), or physical activity treatment/intervention.
* Limited level of oral and written English or Spanish
* Cognitively impaired adults
* Prisoners
* Participants will be excluded from the physical activity and weight loss interventions (but not the smoking cessation component) for:
* Absolute contraindications to exercise (i.e., acute myocardial infarction, complete heart block, acute congestive heart failure, unstable angina, uncontrolled hypertension), metastatic disease or planned elective surgery
* Pregnant or plans to become pregnant.
* Individuals engaging in the physical activity or weight loss interventions must pass pre- physical activity participation screening or obtain medical clearance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Reach/Access | Baseline
  A) We will evaluate the Reach of the risk behavior screening system by assessing the number of cancer survivors exposed to EHR screening and the proportion and representativeness of those who enroll in the study and are randomized. B) We will also evaluate the Reach of the STELLAR intervention by assessing the proportion and representativeness (in terms of disease characteristics, socioeconomic status, telehealth access, technology literacy, race/ethnicity, and insurance status) of those randomized to active intervention who attend at least one treatment session.

SECONDARY OUTCOMES:
Smoking | baseline, 3, 6 and 9 months
  Assessed using Timeline Followback interview, participants who report any smoking, even a puff, in the 7 days prior to the visit will be classified as a person that currently smokes
Body Weight | baseline, 3, 6 and 9 months
  patient reported body weight in lbs.
Self-Reported Weekly Amount (in days and minutes) of Moderate Intensity Physical Activity | baseline, 3, 6 and 9 months
  Patient-reported weekly amount of moderate intensity physical activity in days and minutes will be assessed at each time point. Participants will be asked in the last 7 days, how many days they engaged in moderate intensity activity. Then on the days they were active, about how many minutes they were active (Less than 30 Minutes; 30 minutes to less than 1 hour; 1 hour to less than 1.5 hours; 1.5 hours to less than 2 hours; 2 hours to less than 2.5 hours; Over 2.5 hours)
Godin Leisure Time Exercise Questionnaire | baseline, 3, 6 and 9 months
  It is a valid and reliable measure of PA participation. Participants will indicate frequency of participation in strenuous, moderate, and mild exercise over the past 7 days and average time spent in each activity
Total Healthcare Cost and Amount of Patient Care Utilization | baseline, 3, 6 and 9 months
  The following data will be extracted from the medical record: unplanned, all-cause hospital admissions; potentially avoidable, all-cause emergency department use; 7-day hospital readmissions; and use of triage clinic. Since not all patients receive all their care within the NMHC system, they will also be asked to self-report these data.
Rating of Care Quality as Measured by the Consumer Assessment of Healthcare Providers & Systems Cancer Care Survey) | baseline, 3, 6 and 9 months
  Relevant subscales from AHRQ's Consumer Assessment of Healthcare Providers & Systems (CAHPS) Cancer Care Survey will be used: The specific subscales include:
  1. How Well the Cancer Care Team Communicates with Patients. This subscale asks the participant about provider communication on a 4-point scale from "never" to "always" in terms of how well the provider explained things in an easy-to-understand way, listened carefully to patient, showed respect to patient, and spent enough time with patient.
  2. Availability of Interpreters. This subscale asks yes/no if the patient ever needed an interpreter for visits, and if yes, how often they received one on a 4-point scale from "never" to "always"
  3. Overall Rating of Cancer Team and Cancer Care. This is a single question asking patients to rate their provider on a 1-10 scale with 1 being the worst provider possible and 10 being the best provider possible
Rating of Patient-Provider Communication and Shared Decision-Making as Measured by The Interpersonal Process of Care (IPC32) | baseline, 3, 6 and 9 months
  The Interpersonal Process of Care (IPC32), will assess the patient's thoughts on physician-patient interpersonal interactions. The IPC evaluates:
  1. The patients' assessment of their physician's communication quality by asking how often physicians perform certain activities (e.g. eliciting concerns, explanations) on a scale from 1 = never to 5 = always.
  2. The patient's assessment of how often their provider includes them in decisions about their own health (shared-decision making) on a scale from 1 = never to 5 = always.
  3. The patient's assessment of their provider's interpersonal style based on how often the provider displayed certain behaviors (e.g. compassion, respect) on a scale from 1 = never to 5 = always.
Rating of Symptoms and Functioning as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile | baseline, 3, 6 and 9 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile assesses fatigue, depression, anxiety, ability to participate in social roles and activities, sleep disturbance, physical function, and pain interference/intensity on a 1-5 rating scale with 1 being the worst rating and 5 being the best.
Rating of Quality of Life Using the Health Related Quality of Life Short Form (HRQOL SF-12) | baseline, 3, 6 and 9 months
  Quality of Life will be assessed using the Health Related Quality of Life Short Form (HRQOL SF-12). The tool measures two independent dimensions of HRQOL: physical (physical functioning, role functioning, bodily pain, and general health) and emotional (vitality, social functioning, role functioning and mental health) as well as an aggregate score. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hitsman, PhD, Principal Investigator — Northwestern University; Sofia Garcia, PhD, Principal Investigator — Northwestern University; Siobhan Phillips, PhD, Principal Investigator — Northwestern University; Bonnie Spring, PhD, Principal Investigator — Florida State University
Locations (1):
- Northwestern University-Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data will be made available via a study website. Additionally, the website will contain our intervention manual and materials, templates of all study documents including the protocol, consent form, questionnaires, etc.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available within 1 year of completion of primary data collection
Access Criteria: Please email the principle investigator for access

REFERENCES:
- [Background] Spring B, Garcia SF, Daly E, Jacobs M, Jayeoba M, Jordan N, Kircher S, Kocherginsky M, Mazzetta R, Pollack T, Scanlan L, Scherr C, Hitsman B, Phillips SM. Scalable Telehealth Cancer Care: integrated healthy lifestyle program to live well after cancer treatment. J Natl Cancer Inst Monogr. 2024 Jun 26;2024(64):83-91. doi: 10.1093/jncimonographs/lgae020. PMID 38924795
- [Background] Rendle KA, Tan ASL, Spring B, Bange EM, Lipitz-Snyderman A, Morris MJ, Makarov DV, Daly R, Garcia SF, Hitsman B, Ogedegbe O, Phillips S, Sherman SE, Stetson PD, Vachani A, Wainwright JV, Zullig LL, Bekelman JE. A Framework for Integrating Telehealth Equitably across the cancer care continuum. J Natl Cancer Inst Monogr. 2024 Jun 26;2024(64):92-99. doi: 10.1093/jncimonographs/lgae021. PMID 38924790